CLINICAL TRIAL: NCT02865304
Title: The Efficacy and Safety of Endostar Combined With Taxane-based Regimens for HER-2-negative Metastatic Breast Cancer Patients
Brief Title: The Efficacy and Safety of Endostar Combined With Taxane-based Regimens for HER-2-negative MBC Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FJOC-001
Record Dates: First submitted 2016-05-25; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Angiogenesis; Breast Cancer
Keywords: metastatic breast cancer; HER-2-negative; endostar
MeSH Terms: conditions — Breast Neoplasms | interventions — endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- endostar; taxane (Experimental): Endostar was administered at 7.5 mg/m2, d1-14, q21d and was continued until progressive disease, unacceptable toxicity, consent withdrawal, or completion of 24 months. In the same time,Taxane-based chemotherapy was continued until progressive disease, unacceptable toxicity, consent withdrawal, or up to 8 cycles.
  Interventions: Drug: endostar

INTERVENTIONS:
Drug: endostar

SUMMARY:
The purpose of the present study was to prospectively evaluate the efficacy and safety of endostar, a recombinant product of endostatin, combined with taxane-based regimens for HER-2 negative metastatic breast cancer (MBC) patients.

DETAILED DESCRIPTION:
Endostar is a recombinant product of endostatin, which is an endogenous inhibitor of angiogenesis. Animal studies have shown that endostatin is capable of blocking the proliferation and organization of endothelial cells into new blood vessels in vitro and inhibiting angiogenesis and growth of both primary tumors and secondary metastasis. Regarding breast cancer, in vivo studies showed that the combination of paclitaxel and P125A-endostatin inhibited mammary cancer growth, delayed the onset of multifocal mammary adenocarcinomas, decreased tumor angiogenesis, increased the survival of treated mice in the prevention model, and inhibited lung and lymph node metastasis in the intervention model. Moreover, in a prospective, randomized, controlled, phase II neoadjuvant trial, the combination of rh-endostatin with chemotherapy produced a higher tumor response rate without increasing toxicity in breast cancer patients. Considering these promising data, this prospective study was conducted to evaluate the efficacy and safety of endostar combined with taxane-based regimens for HER-2-negative MBC patients.

ELIGIBILITY:
Inclusion Criteria:

* women with ages between 18-70 years with histologically confirmed MBC documented as HER-2-negative

Exclusion Criteria:

* cannot tolerated chemotherapy
* cardiac insufficiency

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
overall response rate | one year

CONTACTS AND LOCATIONS:
Overall Officials: weiwei huang, doctor, Principal Investigator — Department of Medical Oncology, Fujian Provincial Cancer Hospital, The Teaching Hospital of Fujian Medical University, The Teaching Hospital of Fujian University of Traditional Chinese Medicine, Fuzhou 350014, China

IPD SHARING:
Plan to Share IPD: Undecided